CLINICAL TRIAL: NCT02566772
Title: A Phase 1, Open-Label, Non-Randomized, Safety, Tolerability and Pharmacokinetic Study of TAS3681 in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Study of TAS3681 in Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TO-TAS3681-101; 2015-002745-55 (EudraCT Number)
Record Dates: First submitted 2015-09-25; First posted 2015-10-02 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAS3681 (Experimental): All participants will receive TAS3681 in 28-day cycles. The Escalation phase includes participants who have progressed after abiraterone, enzalutamide and chemotherapy. Eleven dose escalation cohorts are planned, one of which includes a preliminary assessment of food effect. The MTD/recommended dose for further development will be used for participants in the Expansion Phase. The Expansion Phase will enroll participants who have progressed after abiraterone or enzalutamide with chemotherapy consisting of no more than 2 prior taxane-based therapies (Group A) or without any chemotherapy (Group B). Participants receive TAS3681 until discontinuation criteria are met.
  Interventions: Drug: TAS3681

INTERVENTIONS:
Drug: TAS3681 — TAS3681 will be provided as 100 mg tablets to be administered orally in 28-day cycles. The number of cycles is approximately 6, or until discontinuation criteria is met.

SUMMARY:
The purpose of this trial is to investigate the safety and tolerability of TAS3681, to find the maximum tolerated dose (MTD)/recommended dose of TAS3681 (Escalation Phase) and to further evaluate safety and preliminary efficacy of TAS3681 at the MTD/recommended dose (Expansion Phase).

DETAILED DESCRIPTION:
This is a first in human, multinational, Phase 1, open-label study of TAS3681 evaluating safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity in patients with metastatic castration-resistant prostate cancer (mCRPC) for which there is no standard therapy. Eligible participants will be enrolled to evaluate safety and determine the MTD/recommended dose for TAS3681, including a preliminary evaluation of food effect and antitumor activity. The study will be conducted in 2 parts, Dose Escalation (Enrollment closed) and Expansion (Enrollment Closed). Patients who are continuing to receive clinical benefit may receive drug in the extension part of the study after escalation and expansion are completed.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥18 years of age
2. Histological or cytological evidence of metastatic castrate resistant prostate cancer (excluding neuroendocrine differentiation and small cell histology) who are castration resistant and have:

   1. Dose escalation: documented progression defined in PCWG3 and/or intolerance to abiraterone and/or enzalutamide therapy, as well as 1 or more chemotherapies.
   2. Expansion:

   I. Group A: documented progression after abiraterone or enzalutamide and chemotherapy consisting of no more than 2 prior taxane-based therapies

   ii. Group B: documented progression after only abiraterone or enzalutamide therapy without any chemotherapy

   iii. Measurable disease per RECIST 1.1 and/or bone metastases
3. ECOG performance status of ≤1 on Day 1 Cycle 1
4. Ongoing androgen deprivation with serum testosterone <50 ng/dL
5. Expansion Phase only: willingness to undergo baseline core biopsies, if feasible
6. Ability to take medication orally
7. Adequate organ function
8. Agree to use effective contraception during the study and for 30 days after the last dose of TAS3681
9. Willing to comply with scheduled visits and procedures

Exclusion Criteria:

1. QTcF ≥ 450 ms, history of QTc prolongation or predisposition for QTc prolongation or family history of sudden cardiac death or QT prolongation
2. History or presence of heart failure or left ventricular dysfunction with ejection fraction <40% within the previous 6 months; if >6 months cardiac function within normal limits and free of cardiac-related symptoms
3. History or presence of atrial fibrillation, atrial flutter, or paroxysmal supraventricular tachycardia; the presence or history of ventricular arrhythmias including ventricular fibrillation and ventricular tachycardia
4. Presence of cardiac pacemaker or implantable cardioverter-defibrillator
5. History or presence of bradycardia or conduction abnormalities
6. History or presence of cardiac arrest or unexplained syncope
7. Hypokalemia
8. History of myocardial infarction or severe unstable angina
9. Any medication administered within 2 weeks prior to 1st dose of TAS3681 that is known to prolong the QT interval or be arrhythmogenic
10. Received G-CSF, radiotherapy for extended field, anticancer chemotherapy, investigational agents, or major surgery within 4 weeks of study drug administration; receipt of anticoagulant or CYP3A inhibitor within 2 weeks of study drug administration
11. Serious illness or medical condition that could affect the safety or tolerability of study treatments
12. Received prior treatment with TAS3681
13. User of herbal products
14. Any condition or reason that in the opinion of the investigator, interferes with the ability of the participant to participate in the trial
15. To be eligible to participate in the food effect assessment (Escalation Phase only), participants must not have a history or presence of any clinically significant abnormality involving the gastrointestinal tract and an inability to fast for a minimum of 8 hours

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicities | Through 1 month
Escalation Phase: Number of patients with treatment-emergent adverse events and significant ECG abnormalities | Through 6 months (or until patient discontinuation)
  Based on treatment-emergent adverse events, serious adverse events (SAEs), clinical laboratory tests, vital signs, 12-lead electrocardiograms (ECGs)
Expansion Phase: Overall Response Rate (ORR) | Through 6 months (or until patient discontinuation)
  ORR based on investigator-assessed radiographic response per PCWG3/modified RECIST 1.1

SECONDARY OUTCOMES:
Escalation Phase: Prostate Specific Antigen (PSA) response | Up to 6 months (or until patient discontinuation)
Escalation Phase: Time to PSA progression | Up to 6 months (or until patient discontinuation)
Escalation Phase: Maximum concentration of TAS3681 in plasma | Through Day 15 in Cycle 1 (each cycle is 28 days)
Escalation Phase: Time to reach maximum concentration of TAS3681 | At Day 15 in Cycle 1 (each cycle is 28 days)
Escalation Phase: Area under the concentration-time curve of TAS3681 | Through Day 15 in Cycle 1 (each cycle is 28 days)
Escalation Phase: Terminal half-life time of TAS3681 | Through Day 15 in Cycle 1 (each cycle is 28 days)
Escalation Phase: Accumulation ratio of TAS3681 | Through Day 15 in Cycle 1 (each cycle is 28 days)
Escalation Phase: Tumor response per PCWG3/RECIST 1.1 including ORR, and duration of response (DOR) | Through 6 months ( or until patient discontinuation)
Expansion Phase: Prostate Specific Antigen (PSA) response | Up to 6 months (or until patient discontinuation)
Expansion Phase: Number of patients with treatment-emergent adverse events and significant ECG abnormalities | Through 6 months (or until patient discontinuation)
  Based on treatment-emergent adverse events, serious adverse events (SAEs), clinical laboratory tests, vital signs, 12-lead ECGs
Expansion Phase: Maximum concentration of TAS3681 in plasma | Through Day 15 during Cycle 1 (each cycle is 28 days)
Expansion Phase: Time to reach maximum concentration of TAS3681 | Through Day 15 during Cycle 1 (each cycle is 28 days)
Expansion Phase: Area under the concentration-time curve of TAS3681 | Through Day 15 during Cycle 1 (each cycle is 28 days)
Expansion Phase: Terminal half-life time of TAS3681 | Through Day 15 of Cycle 1 (each cycle is 28 days)
Expansion:Tumor response measures including duration of response (DOR), radiologic progression-free survival (rPFS), overall survival (OS), clinical benefit rate (CBR; percentage of participants with complete response, partial response or stable disease) | Through 6 months (or until patient discontinuation)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (11):
  - Univeristy of California Davis Comprehensive Cancer Center, Sacramento, California
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - UMMC-Cancer Center and Research Institute, Jackson, Missouri
  - GU Research Network / Urology Cancer Center, Omaha, Nebraska
  - Premier Oncology Group, Edison, New Jersey
  - MSKCC, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin-Carbone Cancer Center, Madison, Wisconsin
- France (10):
  - Institut Bergonie, Bordeaux
  - Centre Léon BERARD, Lyon
  - Hospices Civils de Lyon, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut régional du Cancer de Montpellier - ICM Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - HEGP- Hôpital Européen Georges Pompidou, Paris
  - Centre eugenie Marquis, Rennes
  - Hopital Foch, Suresnes
  - Gustave Roussy, Villejuif
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala d Oncologia - L Hospitalet de Llobregat, Barcelona
  - Hospital Provincial de Castellon, Castellana
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitari Parc Taulí, Sabadell
  - Hospital Marques de Valdecilla, Santander
- United Kingdom (5):
  - Sarah Cannon Research Institute UK, London, England
  - The Christie NHS Foundation Trust- The Christie Clinic, Manchester, Greater Manchester
  - Royal Marsden Hospital (RMH) NHS Foundation Trust (DDU), Sutton, Surrey
  - Royal Marsden Hospital (RMH) NHS Foundation Trust, Sutton, Surrey
  - Cambridge University Hospitals NHS Foundation, Cambridge

IPD SHARING:
Plan to Share IPD: No